CLINICAL TRIAL: NCT04381195
Title: Relationships, Employment, Autonomy, and Life Satisfaction - #REALSadultlife
Brief Title: Relationships, Employment, Autonomy, and Life Satisfaction (REALS) Study
Acronym: REALS
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Autism Speaks (Other)
Responsible Party: Principal Investigator, Carla Mazefsky, Professor of Psychiatry, University of Pittsburgh
Other Study IDs: STUDY19080355; 11923 (Other Grant/Funding Number: Autism Speaks); R01HD100392 (NIH)
Record Dates: First submitted 2020-05-01; First posted 2020-05-08 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Sound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aim 1: Item Drafting and Revising (Aim 1). Together with a stakeholder panel of autistic adults and adults with IDD and parents/caregivers, the study investigators will generate an item pool based on the conceptual model.
  Interventions: Diagnostic Test: REALS Development
- Aim 2: Item Calibration (Aim 2). Measures will be completed online and therefore the sample will include those with self-reported IDD or autism diagnoses and their caregivers (total n of 1000 each)
  Interventions: Diagnostic Test: REALS Testing

INTERVENTIONS:
Diagnostic Test: REALS Development — Complete drafting of an item pool (adults with ASD, parents, adult service providers); Assign items to all parts of our conceptual framework to ensure sufficient construct coverage across employment, social, and independent living domains; and Conduct cognitive interviews with 25 caregivers of adults with ASD and 25 self-reporting adults with ASD.
  Other Names: Develop and refine an item pool for measuring adult outcomes in ASD
  Groups: Aim 1
Diagnostic Test: REALS Testing — A national sample of proxy reporters (e.g., parents, clinicians, group home staff) for 1000 autistic adults and self-reporting autistic adults and adults with other IDD will complete the REALS draft items and a co-calibration battery to establish psychometrics, generate short-forms, and ensure applicability across adults with ASD.
  Other Names: Derive caregiver and self-report short-forms that are reliable and valid
  Groups: Aim 2

SUMMARY:
One of the major methodological obstacles to more informed policies and programs to support the successful transition to adulthood in autism spectrum disorder (ASD) is the absence of suitable measures of meaningful outcomes for adults. Currently available options include (a) measures designed for children that largely fail to capture concepts pertinent in adulthood or (b) the use of broad, often dichotomous outcomes (e.g., employed or not) that are insufficiently sensitive for monitoring progress. The objective of this project is to develop efficient and validated proxy and self-report measures for autistic adults and adults with other IDD in the domains of relationships, employment, autonomy, and life satisfaction called the REALS.

This study will build on prior success in applying methods from the Patient-Reported Outcomes Measurement Information System (PROMIS®) to measurement development in ASD and will utilize a national sample of 500 autistic adults capable of self-report and 500 caregivers of autistic adults representative of the entire range of speaking level.

DETAILED DESCRIPTION:
A major methodological obstacle to more informed policies to support autistic adults and adults with other intellectual and developmental disabilities (IDD) is the absence of suitable measures of outcomes for autistic adults. Landmark studies of adult outcome have traditionally classified individuals as having good, fair, or poor outcomes, a rating which has low reliability and is generally insensitive to treatment-related changes. Other studies have utilized adaptive behavior scales as functional outcome measures even though they were not designed for that purpose, such as the Vineland Adaptive Behavior Scales (VABS). Importantly, meaningful aspects of adult life are related to, but different than, adaptive function, with the former being the key endpoints of intervention (e.g., employment, friendships) and adaptive function representing important abilities (e.g., communication, ability to follow instructions) that contribute to improved outcomes. Further, the VABS and similar measures were originally developed for children to confirm disability status in school, and as such they have limited coverage of adult content. Therefore, there is an urgent need for sensitive and validated measures of adult outcomes.

The completion of these aims will generate, for the first time, a reliable and valid measure of adulthood functioning in ASD that is efficient and broadly applicable across the full range of speaking ability. The availability of such a measure is essential to inform and evaluate program development, understand individual-level factors associated with outcomes, and ultimately to develop actionable items to improve the transition to adulthood and adult life.

The objective of this project is to develop efficient and validated proxy and self-report measures or autistic adults and adults with other IDD -relationships, employment, autonomy, and life satisfaction called the REALS, and establish the validity of the REALS utilizing state-level service utilization data. This study will build on a previous study's success in applying methods from PROMIS® to measurement development in ASD.

Aim 1. Develop and refine an item pool. The REALS study will:

1. Complete drafting of an item pool with expert input (autistic adults, parents, adult service providers, researchers);
2. Assign items to all parts of the conceptual framework to ensure sufficient construct coverage across employment, social, and independent living domains; and
3. Conduct cognitive interviews with 25 caregivers of autistic adults and adults with other IDD and 25 self-reporting adults.

Aim 2. Establish the psychometrics of the REALS and derive caregiver and self-report short-forms that are reliable and valid. A national sample of proxy reporters (e.g., parents, clinicians, group home staff) for 500 adults with ASD representative of the full range of verbal and intellectual abilities and 500 self-reporting autistic adults will complete the REALS draft items and a co-calibration battery to establish psychometrics, generate short-forms, and ensure applicability across autistic adults.

ELIGIBILITY:
Inclusion Criteria:

Across Aims, inclusion criteria are:

1. adult age, defined as 18+ years old;
2. professional diagnosis of ASD or caregiver of an adult with a professional diagnosis of ASD.

Inclusion criteria for caregivers of adults with ASD will be

1. age 18 years or older;
2. caregiver of an autistic adult with at least weekly contact. For adults who cannot self-report, only caregiver report data on the REALS will be collected.

Exclusion Criteria:

Because the goal is to refine the items and ensure coverage of all relevant constructs, the investigators will seek a broad sample to support generalizability and representativeness (there will be no exclusion criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Autistic adults, parents/caregivers of autistic adults, adults with IDD, parents/caregivers of adults with IDD
Sampling Method: Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Relationships, Employment, Autonomy and Life Satisfaction (REALS) Scale | 5 years
  The completion of these aims will generate, for the first time, a reliable and valid measure of adulthood functioning in ASD that is efficient and broadly applicable across the full range of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Mazefsky, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will occur at two levels:
  1. specific requests to analyze de-identified data from the SQL database and
  2. collaboration with NIH to facilitate de-identified data sharing activities for the National Database for Autism Research (NDAR). The investigators will establish final plans for data sharing procedures that are compliant with NIH policy, the Freedom of Information Act, the DHHS Privacy Rule, HIPPA, and the University of Pittsburgh Institutional Review Board (IRB) regulations and will vet all requests for data.
Time Frame: Data may be shared after study completion and publication.
Access Criteria: The investigators of this study will review and determine which specific requests to analyze de-identified data from the SQL database by other researchers will be shared. Investigators will also share data in collaboration with NIH to facilitate de-identified data sharing activities for the National Database for Autism Research (NDAR).